CLINICAL TRIAL: NCT06826170
Title: HYPOFRACTIONATED STEREOTACTIC RADIOTHERAPY/MULTISESSION RADIOSURGERY (HSFRT/MSRS) in RESIDUAL/ RECURRENT NON SECRETING PITUITARY ADENOMAS an EXPLORATORY STUDY
Brief Title: Hypofractionated Radiosurgery to Treat Residual/recurrent Non Secreting Pituitary Adenoma (HYPOADENO)
Acronym: HYPOADENO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYPO_ADENO
Record Dates: First submitted 2025-01-31; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pituitary Neoplasms; Pituitary Adenoma
Keywords: non functioning pitutary adenoma; radiosurgery; multisession radiosurgery; hypofractionated radiosurgery
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Intervention Model Description: Radiosurgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiosurgery (Experimental): Patients suffering from residual/recurrent non functioning pituitary adenoma wil undergo to hypofractionated radiosurgery
  Interventions: Radiation: hypofractionated radiosurgery

INTERVENTIONS:
Radiation: hypofractionated radiosurgery — The total dose will be 25 Gy, delivered in 5 fractions, in 5 consecutive days

SUMMARY:
Single session stereotactic radiosurgery (SRS) is commonly used for patients with non-functioning adenomas. However the SRS can be limited by the proximity of the tumor with the surrounding critical structures (i.e., the optic chiasm).

The goal of the present prospective phase II trial is to investigate early and early delayed toxicity for cranial nerves and pituitary function after hypofractionated stereotactic radiotherapy/multisession radiosurgery (hSFRT/mSRS) in residual/ recurrent non secreting pituitary adenomas. Secondary end points are late toxicity and tumour growth local control.

All the enrolled patients will undergo radiosurgical treatment with a hypofractionation schedule Following radiotherapy, follow-up will be scheduled every 6 months during the first year post-radiosurgery and then annually, with the same tests.

The baseline examination and the follow-up assessment will include magnetic resonance imaging (MRI), full blood counts and blood chemistry tests, neuro-ophtalmology evaluation, physical and psychological examination that included a quality-of-life (EORTC Quol 30; BN 20) and a Hospital Anxiety and Depression Scale (HADS).

DETAILED DESCRIPTION:
Aims The main aim of our study is to analyze the effect of 5-session hypofractionated radiotherapy/multisession radiosurgery in treating NFAs in terms of toxicity and local control.

Study design This study is an exploratory study: patient's and treatment's data will be prospectively collected in a database and they will then be described and analyzed.

Criteria of analysis

All these points will be recorded and analyzed:

* Local control measured from the date of mSRS until progression or death, censored at the time of last clinical follow-up or imaging.
* Overall survival measured from the date of diagnosis until death, censored at the time of last clinical follow-up or imaging.
* Visual acuity improvement/worsening will be defined by reading increases/decreases equal of 1 or more lines; visual field will be considered improved or worsened for decreases or increase in the extension of the defect area. In order to compare pre- and post-treatment data, the results will be registered.
* Pituitary toxicity will be defined as a clinically relevant reduction compared to the baseline of ACTH, GH, TSH, testosterone in men, period disturbances in women, new onset of diabetes insipidus due to ADH deficiency. Hormonal changes will be defined relevant if a medical therapy change\introduction become mandatory.
* Other treatment-related toxicity based on CTCAE v4.0.
* Presence of adverse events based on CTCAE v4.0.
* Quality of life evaluated by "Quality of life EORTC - QLQ C30 and BN20" and "Hospital Anxiety and Depression Scale (HADS)". (25-28) (Appendix 1 and 2)

Study population Patients suffering from recurrent/residual non secreting pituitary adenoma. Twenty-five patients will be enrolled.

Study treatment Patients will receive hSFRT/mSRS in 5 consecutive days over 7 elapsed days, with extension over a weekend allowed.

Radiation treatment features Following sub-total surgery or in case of progressive disease patients will be enrolled and a CT and MRI simulation will be performed. A treatment for hypofractionated stereotactic radiotherapy/multifraction radiosurgery (hSHRT/mSRS) will be planned. The planning tumor volume (PTV) will be the residual/recurrent tumor + 0-2 mm as defined on the MRI images. To better define the tumor volume T1 with and without contrast enhancement, with and without fat saturation and T2 axial voloumetric sequences will be acquired and then fused. The prescription isodose line will cover at least 95% of the PTV; undercoverage to 90% will be allowed near organs at risk. Normal organ dose constraints will be 98% of the optic pathways receiving less than 27.5 Gy and brainstem maximum point dose of 30 Gy in 5 fractions, undercovering the PTV to meet these limits.

Patient Assessment and Outcome Reporting The baseline examination will include simulation CT and magnetic resonance imaging (MRI), thereafter full blood counts and blood chemistry tests, neuro-ophtalmology evaluation, physical and psychological examination that included a quality-of-life (EORTC Quol 30; BN 20) and a Hospital Anxiety and Depression Scale (HADS).

Following radiotherapy, follow-up will be scheduled every 6 months during the first year post-radiosurgery and then annually, with the same tests.

Tumor progression will be defined according to the modified WHO criteria as an increase in tumor size by 25 percent. Consensus between the two examining radiologists will be achieved if the target lesions selected differed between the two radiologists. In case of tumor progression, patients will be treated at the investigators' discretion.

Toxicity and adverse events will be graded according to the National Cancer Institute Common Toxicity Criteria, version 4.0, with a score of 1 indicating mild adverse effects, a score of 2 moderate adverse effects, a score of 3 severe adverse effects, and a score of 4 life-threatening adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Residual or progressive non secreting pituitary adenoma;
* Exclusion of other treatment approach (second surgery, wait and scan; suppressive therapy) by a multidisciplinary team
* Age ≥ 18 years; KPS ≥ 70
* Written privacy consent;
* Ability to give informed consent;

Exclusion Criteria:

* Previous cranial irradiation;
* Diagnosis of secreting adenoma;
* pregnancy status;
* unable to undergo MRI or CT scans;
* unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Early and late treatment related toxicity | From the treatment to 36th month post-treatment
  - Treatment-related toxicity based on CTCAE v4.0.
Impact of the treatment on visual acuity | From the treatment time to the 36th month post-treatment
  - Visual acuity (VA) improvement/worsening will be defined by reading increases/decreases equal of 1 or more lines (Vdetermined by the best performance on the Snellen Chart).
Impact of the treatment on the visual field | From the treatment time to the 36th month post-treatment
  The visual field (VF) is a continuous quantitative variable described by the mean deviation (VFMD) value, which is a summary measure of vision average loss across the visual field. VFMD values at follow-up visits that are less negative than the baseline are considered an improvement, while more negative values are considered a worsening.
Impact of the treatment on the pituitary function | From the treatment time to the 36th month post-treatment
  Pituitary toxicity will be defined as a clinically relevant reduction compared to the baseline of ACTH, GH, TSH, testosterone in men, period disturbances in women, new onset of diabetes insipidus due to ADH deficiency. Hormonal changes will be defined relevant if a medical therapy change\introduction become mandatory.

SECONDARY OUTCOMES:
Tumor control | From the treatment time to the 36th month post-treatment
  Tumor progression will be defined according to the modified WHO criteria as an increase in tumor size by 25 percent
Impact of the treatment on the quality of life | From the treatment time to the 36th month post-treatment.
  Quality of life will be evaluated acoording to Quality of life (EORTC QLQ C30 - QLQ BN 20) variations
Impact of the treatment on anxiety and depression | From the treatment time to the 36th month post-treatment
  Anxiety and Depression experienced by the patients will be evaluated according to "Hospital Anxiety and Depression Scale (HADS)" variations.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico C Besta, Milan, Milan, Italy